CLINICAL TRIAL: NCT03475706
Title: A Phase 2b, Multicenter, Randomized, Double-Blind, Placebo-Controlled, Parallel-Group Study to Evaluate the Efficacy and Safety of Oral Solabegron Immediate Release Tablets in the Treatment of Overactive Bladder (OAB) in Adult Female Subjects
Brief Title: Evaluation of the Efficacy and Safety of Solabegron Tablets for Treatment of Overactive Bladder in Adult Women
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Velicept Therapeutics, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: VEL-2002
Record Dates: First submitted 2018-03-12; First posted 2018-03-23 (Actual); Last update posted 2020-03-02 (Actual); Status verified 2019-01

CONDITIONS: Overactive Bladder
Keywords: overactive bladder; urinary conditions; urgency urinary incontinence; urgency; micturitions
MeSH Terms: conditions — Urinary Bladder, Overactive | interventions — solabegron

STUDY DESIGN:
Intervention Model Description: This is a Phase 2b, multicenter, randomized, double-blind, placebo-controlled, parallel-group study. Eligible female subjects (N=406) with symptoms of overactive bladder for at least 6 months will enter a 14-day single-blind Run-in Period. Subjects (N=375) who meet prespecified criteria based on data entered into an electronic diary over 3 days will be randomized 1:1:1 (125 subjects per arm) to receive solabegron immediate release tablets, low dose or high dose, or matching placebo.
Who Masked: Participant, Investigator
Masking Description: Sponsor representatives Site monitors Data managers Statisticians
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- Solabegron immediate release tablets low dose (Experimental)
  Interventions: Drug: Solabegron immediate release tablets, low dose
- Solabegron immediate release tablets high dose (Experimental)
  Interventions: Drug: Solabegron immediate release tablets, high dose
- Placebo Comparator (Placebo Comparator)
  Interventions: Drug: Matching Placebo

INTERVENTIONS:
Drug: Solabegron immediate release tablets, low dose — twice daily for 12 weeks.
  Arms: Solabegron immediate release tablets low dose
Drug: Solabegron immediate release tablets, high dose — twice daily for 12 weeks.
  Arms: Solabegron immediate release tablets high dose
Drug: Matching Placebo — twice daily for 12 weeks.
  Arms: Placebo Comparator

SUMMARY:
This is a Phase 2b, multicenter, randomized, double-blind, placebo-controlled, parallel-group study designed to evaluate the efficacy, safety, and tolerability of solabegron immediate release low dose or high dose tablets, compared to matched placebo, administered twice daily for 12 weeks to adult female subjects with overactive bladder symptoms (frequency, urgency, and predominantly urgency incontinence) for at least 6 months.

ELIGIBILITY:
Inclusion Criteria:

* Adult female subjects 18 to 80 years of age, with a ≥ 6-month history of symptoms of overactive bladder including: frequency, urgency, and urgency urinary incontinence. Subjects must provide written informed consent and either be of non-childbearing potential or of childbearing potential meeting specific criteria (e.g., negative pregnancy test, sexual inactivity, acceptable methods of birth control, and use of hormonal contraceptives).

Exclusion Criteria:

* Subjects must have no history of pelvic or bladder disease, e.g., Grade 3/4 uterine prolapse, urogenital malignancy within the past 2 years, surgery for stress incontinence or pelvic prolapse repair within the past 6 months, or bladder injections with botulinum toxin at any time.
* Diabetes insipidus or poorly controlled Type 1 or Type 2 diabetes mellitus
* Cardiac conditions: prior cardiovascular events or procedures within 6 months of screening; congestive heart failure; abnormal ECG findings, including ECG QT correction interval (QTc) > 470 msec at the Screening Visit; systolic blood pressure ≥ 180 mmHg or diastolic blood pressure ≥100mmHg, or heart rate > 100 beats per minute.
* Abnormal tests of liver function
* History of prior infection due to HIV or hepatitis B or hepatitis C virus
* Allergy or hypersensitivity to solabegron or mirabegron
* Women of childbearing potential: breastfeeding, pregnant, or actively trying to become pregnant
* Participation in a trial of an investigational or marketed drug ≤ 30 days prior to the Screening Visit or in any clinical trial of an investigational drug that may affect urinary function within 3 months prior to Screening Visit.
* Inability to read, understand, or complete study-related materials.

Ages: 18 Years to 80 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 438 (Actual)
Dates: Start 2018-02-19 (Actual); Primary Completion 2019-01-24 (Actual); Study Completion 2019-01-30 (Actual)

PRIMARY OUTCOMES:
Change from Baseline in mean number of micturitions per 24h at Week 12 | Micturitions will be assessed prior to randomization and at Week 12 (Visit 6).
  Micturition events will be recorded by subjects in an eDiary using a smartphone device during 3-day diary periods prior to randomization and at 12 weeks.

SECONDARY OUTCOMES:
Urinary Incontinence (1) | Prior to Randomization (Baseline) and at Weeks 4, 8, and 12
  Change from Baseline in mean number of urgency urinary incontinence episodes per 24h.
Urinary Incontinence (2) | Prior to Randomization (Baseline) and at Weeks 4 and 8
  Percentage change from Baseline in mean number of urgency urinary incontinence episodes per 24h.
Urinary Incontinence (3) | Prior to Randomization (Baseline) and at Weeks 4, 8, and 12
  Proportion of subjects with no episodes of urgency urinary incontinence per 24h.
Urinary Incontinence (4) | Prior to Randomization (Baseline) and at Weeks 4, 8, and 12
  Proportion of subjects with no episodes of urinary incontinence (urgency or non-urgency) per 24h.
Urinary Incontinence (5) | Prior to Randomization (Baseline) and at Weeks 4, 8, and 12
  Change from Baseline in total urinary incontinence episodes (urgency and non-urgency) per 24h.
Micturitions (1) | Prior to Randomization (Baseline) and at Weeks 4 and 8
  Change from Baseline in mean number of micturitions per 24h.
Micturitions (2) | Prior to Randomization (Baseline) and at Weeks 4, 8, and 12
  Percentage change from Baseline in mean number of micturitions per 24h.
Micturitions (3) | Prior to Randomization (Baseline) and at Weeks 4, 8, and 12
  Percentage of subjects with <8 micturitions per 24h.
Micturitions (4) | Prior to Randomization (Baseline) and at Weeks 4, 8, and 12
  Change from Baseline in mean number of nocturnal voids per 24h.
Urine Void Volume (1) | Prior to Randomization (Baseline) and at Weeks 4, 8, and 12
  Change from Baseline in average void volume over 24h.
Urine Void Volume (2) | Prior to Randomization (Baseline) and at Weeks 4, 8, and 12
  Percentage change from Baseline in average void volume over 24h.
Urine Void Volume (3) | Prior to Randomization (Baseline) and at Weeks 4, 8, and 12
  Change from Baseline in maximum individual void volume over 24h.
Urine Void Volume (4) | Prior to Randomization (Baseline) and at Weeks 4, 8, and 12
  Percentage change from Baseline in maximum individual void volume over 24h.
Urgency (1) | Prior to Randomization (Baseline) and at Weeks 4, 8, and 12
  Proportion of subjects with urges with a mean grade of 3 or 4 per 24h.
Urgency (2) | Prior to Randomization (Baseline) and at Weeks 4, 8, and 12
  Change from Baseline in urgency assessments per 24h associated with micturitions and incontinence.
Patient Reported Outcomes (1) | Prior to Randomization (Baseline) and at Weeks 4, 8, and 12
  Patient Perception of Bladder Condition
Patient Reported Outcomes (2) | Prior to Randomization (Baseline) and at Weeks 4, 8, and 12
  Change from Baseline in Symptom Bother Score (OAB-q short form).
Patient Reported Outcomes (3) | Prior to Randomization (Baseline) and at Weeks 4, 8, and 12
  Change from Baseline in health-related quality of life (OAB-q short form).

CONTACTS AND LOCATIONS:
Locations (80):
- United States (80):
  - Velicept Investigative Site - Birmingham, Birmingham, Alabama
  - Velicept Investigative Site - Gulf Shores, Gulf Shores, Alabama
  - Velicept Investigative Site - Mobile, Mobile, Alabama
  - Velicept Investigative Site - Tempe, Tempe, Arizona
  - Velicept Investigative Site - Tucson, Tucson, Arizona
  - Velicept Investigative Site - Little Rock, Little Rock, Arkansas
  - Velicept Investigative Site - Anaheim, Anaheim, California
  - Velicept Investigative Site - Arcadia, Arcadia, California
  - Velicept Investigative Site - Canoga Park, Canoga Park, California
  - Velicept Investigative Site - Huntington Beach, Huntington Beach, California
  - Velicept Investigative Site - Los Alamitos, Los Alamitos, California
  - Velicept Investigative Site - Los Angeles, Los Angeles, California
  - Velicept Investigative Site - Norco, Norco, California
  - Velicept Investigative Site - Sacramento, Sacramento, California
  - Velicept Investigative Site - San Diego, San Diego, California
  - Velicept Investigative Site - San Marcos, San Marcos, California
  - Velicept Investigative Site - Thousand Oaks, Thousand Oaks, California
  - Velicept Investigative Site - Denver, Denver, Colorado
  - Velicept Investigative Site - Waterbury, Waterbury, Connecticut
  - Velicept Investigative Site - Clearwater, Clearwater, Florida
  - Velicept Investigative Site - Deland, DeLand, Florida
  - Velicept Investigative Site - Doral, Doral, Florida
  - Velicept Investigative Site - Jupiter, Jupiter, Florida
  - Velicept Investigative Site - Lake City, Lake City, Florida
  - Velicept Investigative Site - Miami, Miami, Florida
  - Velicept Investigative Site - Ponte Vedra, Ponte Vedra, Florida
  - Velicept Investigative Site - Port St Lucie, Port Saint Lucie, Florida
  - Velicept Investigative Site - West Palm Beach, West Palm Beach, Florida
  - Velicept Investigative Site - Winter Haven, Winter Haven, Florida
  - Velicept Investigative Site - Marietta, Marietta, Georgia
  - Velicept Investigative Site - Blackfoot, Blackfoot, Idaho
  - Velicept Investigative Site - Meridian, Meridian, Idaho
  - Velicept Investigative Site - Wauconda, Wauconda, Illinois
  - Velicept Investigative Site - Elwood, Elwood, Indiana
  - Velicept Investigative Site - Evansville, Evansville, Indiana
  - Velicept Investigative Site - Newton, Newton, Kansas
  - Velicept Investigative Site - Louisville, Louisville, Kentucky
  - Velicept Investigative Site - Metairie, Metairie, Louisiana
  - Velicept Investigative Site - New Orleans, New Orleans, Louisiana
  - Velicept Investigative Site - Shreveport, Shreveport, Louisiana
  - Velicept Investigative Site - Boston, Boston, Massachusetts
  - Velicept Investigative Site - New Bedford, New Bedford, Massachusetts
  - Velicept Investigative Site - North Attleborro, North Attleboro, Massachusetts
  - Velicept Investigative Site - Watertown, Watertown, Massachusetts
  - Velicept Investigative Site - Kalamazoo, Kalamazoo, Michigan
  - Velicept Investigative Site - St. Louis, St Louis, Missouri
  - Velicept Investigative Site - Omaha, Omaha, Nebraska
  - Velicept Investigative Site - Las Vegas, Las Vegas, Nevada
  - Velicept Investigative Site - Brick, Brick, New Jersey
  - Velicept Investigative Site - Vorhees, Voorhees Township, New Jersey
  - Velicept Investigative Site - Albuquerque, Albuquerque, New Mexico
  - Velicept Investigative Site - New York, New York, New York
  - Velicept Investigative Site - Williamsville, Williamsville, New York
  - Velicept Investigative Site - Charlotte, Charlotte, North Carolina
  - Velicept Investigative Site - Wilmington, Wilmington, North Carolina
  - Velicept Investigative Site - Winston-Salem, Winston-Salem, North Carolina
  - Velicept Investigative Site - Cincinnati, Cincinnati, Ohio
  - Velicept Investigative Site - Cleveland, Cleveland, Ohio
  - Velicept Investigative Site - Columbus, Columbus, Ohio
  - Velicept Investigative Site - Marion, Marion, Ohio
  - Velicept Investigative Site - Middleburg Heights, Middleburg Heights, Ohio
  - Velicept Investigative Site - Warwick, Warwick, Rhode Island
  - Velicept Investigative Site - Mt. Pleasant, Mt. Pleasant, South Carolina
  - Velicept Investigative Site - Myrtle Beach, Myrtle Beach, South Carolina
  - Velicept Investigative Site - Jackson, Jackson, Tennessee
  - Velicept Investigative Site - Knoxville, Knoxville, Tennessee
  - Velicept Investigative Site - Nashville, Nashville, Tennessee
  - Velicept Investigative Site - Austin, Austin, Texas
  - Velicept Investigative Site - Beaumont, Beaumont, Texas
  - Velicept Investigative Site - Lampasas, Lampasas, Texas
  - Velicept Investigative Site - Longview, Longview, Texas
  - Velicept Investigative Site - San Antonio, San Antonio, Texas
  - Velicept Investigative Site - Clinton, Clinton, Utah
  - Velicept Investigative Site - Salt Lake City, Salt Lake City, Utah
  - Velicept Investigative Site - St. George, St. George, Utah
  - Velicept Investigative Site - West Jordan, West Jordan, Utah
  - Velicept Investigative Site - Newport News, Newport News, Virginia
  - Velicept Investigative Site - Norfolk, Norfolk, Virginia
  - Velicept Investigative Site - Tacoma, Tacoma, Washington
  - Velicept Investigative Site - Kenosha, Kenosha, Wisconsin

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Ohlstein EH, von Keitz A, Michel MC. A multicenter, double-blind, randomized, placebo-controlled trial of the beta3-adrenoceptor agonist solabegron for overactive bladder. Eur Urol. 2012 Nov;62(5):834-40. doi: 10.1016/j.eururo.2012.05.053. Epub 2012 Jun 5. PMID 22695239